CLINICAL TRIAL: NCT05210023
Title: Effect of a Nutrigenetic Intervention on Blood Lipid Markers and Body Composition of Adults With Overweight and Obesity
Brief Title: Nutrigenetic Intervention on Blood Lipid Markers and Body Composition of Adults With Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Tecnológico y de Estudios Superiores de Occidente (Other)
Collaborators: Instituto Tecnológico de Tepic (Unknown); University of Guadalajara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUTRIGENETIC_INTERV07
Record Dates: First submitted 2021-12-31; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Dyslipidemias; Overweight and Obesity
Keywords: nutrigenetic; polymorphisms; dietetic intervention; lipid levels
MeSH Terms: conditions — Dyslipidemias; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, parallel, with 2 study groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrigenetic Diet Group (Experimental): Participants randomly included in this group will receive nutrigenetic menus, i.e., considering the genotypes of the 11 variants analyzed.
  Interventions: Other: NUTRIGENETIC DIET INTERVENTION
- Conventional Diet Group (Experimental): Participants randomly included in this group will receive menus prepared following the international conventional guidelines set out by the WHO, AHA and Official Mexican Standards (NOM) for the treatment of obesity and dyslipidemia.
  Interventions: Other: CONVENTIONAL DIET INTERVENTION

INTERVENTIONS:
Other: NUTRIGENETIC DIET INTERVENTION — Weekly, personalized meal plans (menus) will be provided, prepared based on the anthropometric needs of the patients, with a caloric reduction (-500 kcal). These weekly menus (Sunday to Monday) consist of 5 meal times (breakfast, snack, lunch, snack and dinner). The distribution of the macronutrients: carbohydrates, proteins and fats, as well as the percentages of polyunsaturated, monounsaturated and saturated fatty acids, will be established according to certain nutrigenetic recommendations identified in the reference bibliography.
  Participants included in this group will receive remote (virtual) nutritional counseling every 15 days.
  Other Names: Nutrigenetic diet group
  Arms: Nutrigenetic Diet Group
Other: CONVENTIONAL DIET INTERVENTION — Weekly, personalized meal plans (menus) will be provided, prepared based on the anthropometric needs of the patients, with a caloric reduction (-500 kcal). These weekly menus (Sunday to Monday) consist of 5 meal times (breakfast, snack, lunch, snack and dinner). The distribution of the macronutrients: carbohydrates, proteins and fats, as well as the percentages of polyunsaturated, monounsaturated and saturated fatty acids, will be in accordance with the recommendations made by the WHO (World Health Organization), the AHA (American heart association) and the NOM (Official Mexican Standards) for the treatment of obesity and dyslipidemias.
  Participants included in this group will receive remote (virtual) nutritional counseling every 15 days.
  Other Names: Conventional diet group
  Arms: Conventional Diet Group

SUMMARY:
Obesity is defined as the accumulation of excessive fat, attributed to the maintenance of a positive energy imbalance between calorie intake and expenditure. Obesity contributes to the development of many comorbidities such as type 2 diabetes, cardiovascular diseases, hypertension, metabolic syndrome, and dyslipidemias, among others. Dyslipidemias indicate a high concentration of lipids in the blood. Dyslipidemias cause more than 4 million premature deaths per year.

The pathogenesis of obesity is complex as it involves environmental, sociocultural, physiological, medical, behavioral, genetic, epigenetic, and many other factors. On the other hand, the causes of dyslipidemias can be: genetic / hereditary (primary dyslipidemias) or an inadequate lifestyle (secondary dyslipidemias).

Sufficient evidence indicates that lifestyle, mainly diet, plays a decisive role in the development of diseases such as obesity and dyslipidemias, in addition to that, recent research shows the importance of individual genetic predisposition to suffer from diseases. Data based on genome-wide association studies suggest a genetic predisposition for obesity and dyslipidemias with identification of various genes and genetic variations associated with these conditions. In this sense, the postulates of nutrigenetics as applied science are emphasized, since it states that food components can act on the human genome, directly or indirectly, to alter the expression of genes and gene products; diet can potentially compensate or accentuate the effects of genetic polymorphisms; and the consequences of a certain diet depend on the balance of health and disease states and the genetic background of an individual.

Therefore, when advising a change in diet and lifestyle as prevention and as part of the treatment for obesity and dyslipidemias, it is considered that a nutrigenetic intervention, that is, the administration of a diet designed according to genotypic characteristics and personal phenotypic, will have a much greater positive impact on the health status of people with detected genetic variations that make them susceptible to these pathologies.

For this reason, the implementation of nutrigenetic interventions could be a timely and successful avant-garde treatment to mitigate various cardiometabolic diseases such as dyslipidemias and others that are highly prevalent worldwide.

DETAILED DESCRIPTION:
After the selection of the population, the patients undergo a molecular diagnosis: DNA will be extracted from peripheral blood with the High Pure PCR (Polymerase Chain Reaction) Template Preparation Kit (Roche). Then certain polymorphisms will be determined by allelic discrimination with TaqMan® probes with real-time PCR.

The polymorphisms under study will be the following:

ABCA1 (ATP-binding cassette transporter ABCA1) rs9282541 PPARG (Peroxisome Proliferator Activated Receptor Gamma) rs1801282 LIPC (hepatic lipase) rs1800588 CETP (Cholesteryl ester transfer protein) rs708272 LPL (Lipoprotein lipase) rs13702 FABP2 (fatty acid binding protein 2) rs1799883 APOA5 (Apolipoprotein A-V) rs662799 APOC3 (Apolipoprotein C-III) rs5128 APOA1 (Apolipoprotein A-I) rs670 APOE (Apolipoprotein E) rs429358 and rs7412

Patients will be randomized into two different treatment groups. Randomization will be stratified according to age, BMI and sex. The allocation ratio will be 1: 1 and parallel intervention.Then, trained nutritionists will deliver the intervention according to the patient group and they will be followed-up for 8 weeks, which includes 3 face-to-face evaluations (baseline, 1st month and final) and 5 remote consultations, via zoom, every 15 days

Interventions will be provided as follows:

NUTRIGENETIC DIET INTERVENTION Weekly, personalized meal plans (menus) will be provided, prepared based on the anthropometric needs of the patients, with a caloric reduction (-500 kcal). These weekly menus (Sunday to Monday) consist of 5 meal times (breakfast, snack, lunch, snack and dinner). The distribution of the macronutrients: carbohydrates, proteins and fats, as well as the percentages of polyunsaturated, monounsaturated and saturated fatty acids, will be established according to certain nutrigenetic recommendations identified in the reference bibliography.

CONVENTIONAL DIET INTERVENTION Weekly, personalized meal plans (menus) will be provided, prepared based on the anthropometric needs of the patients, with a caloric reduction (-500 kcal). These weekly menus (Sunday to Monday) consist of 5 meal times (breakfast, snack, lunch, snack and dinner). The distribution of the macronutrients: carbohydrates, proteins and fats, as well as the percentages of polyunsaturated, monounsaturated and saturated fatty acids, will be in accordance with the recommendations made by the WHO (World Health Organization), the AHA (American Heart Association) and the NOM (Official Mexican Standards) for the treatment of obesity and dyslipidemias

The 3 face-to-face evaluations (baseline, 1st month, final) will include anthropometric and biochemical evaluations. Therefore, the following criteria will be measured:

Weight (kg) Height (cm) BMI(kg/m2) Waist circumference and hip circumference (cm) Blood pressure Body composition determination

Blood will be obtained from the antecubital vein, it will be centrifuged to obtain the serum and later it will determine:

Glucose (mg / dL) Total cholesterol (mg / dL) Triglycerides (mg / dL) HDL-c (mg / dL) LDL-c (mg / dL) VLDL-c (mg / dL) Insulin (microIU/mL) C-reactive protein (mg/L) Interleukins, among other parameters

Every 15 days there will be virtual remote consultations, through the zoom platform. In these sessions, the nutritional clinical history and various medical and dietary questionnaires will be applied to evaluate secondary results. In addition, a new food plan will be delivered, according to the needs of the participant and taking into account the characteristics of the experimental treatment to which they belong.

This research will be conducted at The Institute of Translational Nutrigenetics and Nutrigenomics, Department of Molecular Biology and Genomics, Health Sciences University Center, University of Guadalajara, Guadalajara, Mexico

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-50 years old
* Mexican- Mexican ancestry (3 generations)
* Live in Guadalajara, Jalisco or metropolitan area.
* Being overweight or obese BMI 25> 40
* Waist circumference:

Women> 80 cm, Men> 94 cm.

-Availability to attend virtual nutritional consultations

Exclusion Criteria:

* Not meeting the inclusion criteria.
* Pregnancy or breastfeeding
* Gastrointestinal disorders
* Endocrinopathies
* Cardiovascular events
* Diagnosed psychiatric illnesses.
* Diagnosed diabetes
* Take lipid-lowering drugs
* Autoimmune diseases.
* Covid +

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Lipid profile change | Baseline, week 4, week 8
  Measurements of total cholesterol, LDL cholesterol, VLDL cholesterol, HDL cholesterol, and triglycerides will be evaluated to assess lipid profile change.

SECONDARY OUTCOMES:
Body composition change | Baseline, week 4, week 8
  Body fat mass (% BFM), body fat percentage (%BF) and skeletal muscle mass (% SMM) will be evaluated to assess body composition change. Measurements will be assessed using multifrequency bioelectrical impedance analysis (BIA)
Visceral fat index change | Baseline, week 4, week 8
  Visceral fat index change will be evaluated to assess body composition change and fat loss. Measurement will be assessed using multifrequency bioelectrical impedance analysis (BIA)
Body Weight change | Baseline, week 4, week 8
  Measurement of body weight (kg) will be evaluated to assess anthropometric change.
Anthropometric measurements change | Baseline, week 4, week 8
  Waist circumference (cm) and hip circumference (cm) will be evaluated to assess anthropometric change.
Body Mass Index (BMI) change | Baseline, week 4, week 8
  Body Mass Index (BMI) allows the identification of overweight and obesity in adults. Weight and height will be combined to report BMI in (kg/m^2)
tumor Necrosis factor- alfa (TNF-alfa) | Baseline, week 4, week 8
  Change in TNF-alfa (pg/ml) will be evaluated as a marker of inflammation
C-reactive protein (CRP) | Baseline, week 4, week 8
  Change in C-reactive protein (CRP)( mg/L) will be evaluated as a marker of inflammation
Interleukins levels | Baseline, week 4, week 8
  Determination of serum levels of Interleukin (IL) 6, IL1, IL10 (pg/ml) will be evaluated as a markers of inflammation
Change in glucose | Baseline, week 4, week 8
  Measuring glucose levels will determine changes in this parameter
Change in blood pressure | Baseline, week 4, week 8
  Systolic and diastolic pressure measurement will determine changes in blood pressure
Adherence to nutritional intervention | Week 4, week 8
  It will be evaluated through changes in food consumption (food frequency questionnaire)
Change in food intake | Baseline, Week 4, week 8
  Change in food intake using Food Frequency Questionnaire
Change in physical activity practice | Baseline, week 8
  Change in physical activity practice using International Physical Activity Questionnaire - Short Form
Change in insulin level | Baseline, week 4, week 8
  Measurement of insulin levels will determine changes in this parameter (microIU/ml)
Insulin Resistance (HOMA-IR) | Baseline, week 4, week 8
  Insulin resistance will be determined using HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) fasting serum glucose (mg/dL) x insulin (mIU /L) / 405

CONTACTS AND LOCATIONS:
Overall Officials: Edgar J Mendivil, PhD, Study Director — Instituto Tecnológico y de Estudios Superiores de Occidente
Locations (1):
- Institute of Translational Nutrigenetics and Nutrigenomics, Department of Molecular Biology and Genomics, Health Sciences University Center, University of Guadalajara,, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
All information provided by participant is strictly confidential, will be used only by the project's research team and will not be available for any other purpose. The results obtained from this study will be published for scientific purposes but the confidentiality of the participants will never be violated. The information or evidence obtained will be eliminated after fulfilling the scientific purposes for which this intervention was proposed.

REFERENCES:
- [Background] Barrea L, Annunziata G, Bordoni L, Muscogiuri G, Colao A, Savastano S; Obesity Programs of nutrition, Education, Research and Assessment (OPERA) Group. Nutrigenetics-personalized nutrition in obesity and cardiovascular diseases. Int J Obes Suppl. 2020 Jul;10(1):1-13. doi: 10.1038/s41367-020-0014-4. Epub 2020 Jul 20. PMID 32714508
- [Background] Corella D, Ordovas JM. Interactions between dietary n-3 fatty acids and genetic variants and risk of disease. Br J Nutr. 2012 Jun;107 Suppl 2(0 2):S271-83. doi: 10.1017/S0007114512001651. PMID 22591901
- [Background] de Luis D, Izaola O, Primo D, Aller R. Role of rs670 variant of APOA1 gene on metabolic response after a high fat vs. a low fat hypocaloric diets in obese human subjects. J Diabetes Complications. 2019 Mar;33(3):249-254. doi: 10.1016/j.jdiacomp.2018.10.015. Epub 2018 Nov 3. PMID 30467071
- [Background] Fall T, Mendelson M, Speliotes EK. Recent Advances in Human Genetics and Epigenetics of Adiposity: Pathway to Precision Medicine? Gastroenterology. 2017 May;152(7):1695-1706. doi: 10.1053/j.gastro.2017.01.054. Epub 2017 Feb 15. PMID 28214526
- [Background] Hannon BA, Khan NA, Teran-Garcia M. Nutrigenetic Contributions to Dyslipidemia: A Focus on Physiologically Relevant Pathways of Lipid and Lipoprotein Metabolism. Nutrients. 2018 Oct 2;10(10):1404. doi: 10.3390/nu10101404. PMID 30279335
- [Background] Sanchez-Moreno C, Ordovas JM, Smith CE, Baraza JC, Lee YC, Garaulet M. APOA5 gene variation interacts with dietary fat intake to modulate obesity and circulating triglycerides in a Mediterranean population. J Nutr. 2011 Mar;141(3):380-5. doi: 10.3945/jn.110.130344. Epub 2011 Jan 5. PMID 21209257
- [Background] Xu M, Ng SS, Bray GA, Ryan DH, Sacks FM, Ning G, Qi L. Dietary Fat Intake Modifies the Effect of a Common Variant in the LIPC Gene on Changes in Serum Lipid Concentrations during a Long-Term Weight-Loss Intervention Trial. J Nutr. 2015 Jun;145(6):1289-94. doi: 10.3945/jn.115.212514. Epub 2015 Apr 29. PMID 25926410
- [Background] Zhang X, Qi Q, Bray GA, Hu FB, Sacks FM, Qi L. APOA5 genotype modulates 2-y changes in lipid profile in response to weight-loss diet intervention: the Pounds Lost Trial. Am J Clin Nutr. 2012 Oct;96(4):917-22. doi: 10.3945/ajcn.112.040907. Epub 2012 Aug 22. PMID 22914552
- [Result] AlSaleh A, O'Dell SD, Frost GS, Griffin BA, Lovegrove JA, Jebb SA, Sanders TAB. Interaction of PPARG Pro12Ala with dietary fat influences plasma lipids in subjects at cardiometabolic risk. J Lipid Res. 2011 Dec;52(12):2298-2303. doi: 10.1194/jlr.P019281. Epub 2011 Sep 23. PMID 21949049

DOCUMENTS (3):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05210023/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05210023/SAP_001.pdf
  • Informed Consent Form (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT05210023/ICF_002.pdf